CLINICAL TRIAL: NCT06955923
Title: Trigger Point Injection in Reducing Pain Following Total Knee Arthroplasty
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: David Grant U.S. Air Force Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FDG20240079H
Record Dates: First submitted 2025-04-25; First posted 2025-05-02 (Actual); Results first posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Trigger Point Pain, Myofascial
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental group - participants receiving trigger point injections (Experimental): The participant will receive trigger point injections with 1% lidocaine without epinephrine in two muscles in the thigh and two muscles in the calf immediately after having knee replacement surgery.
  Interventions: Drug: Trigger point injection (lidocaine)
- Sham comparator - Participants not receiving trigger point injections (Sham Comparator): The patient will not receive an injection, but instead a façade of an injection by having the same physical set-up to prepare for an injection (the same as for the experimental group), but there will be a barrier between the patient's view and the syringe so that he/she will not know an injection was not given.
  Interventions: Other: Sham Comparator

INTERVENTIONS:
Drug: Trigger point injection (lidocaine) — A trigger point injection utilizing lidocaine 1% without epinephrine will be injected into several muscles bellies immediately following surgery to halt a trigger point from forming. One group will receive this type of intervention and the sham group will not receive any type of injection.
  Arms: Experimental group - participants receiving trigger point injections
Other: Sham Comparator — This arm of the study will not receive any injection.
  Arms: Sham comparator - Participants not receiving trigger point injections

SUMMARY:
This study will evaluate the ability of trigger point injections completed immediately following a total knee arthroplasty decrease pain scores and opioid use compared to sham injections. Given the current state of opioid dependency in the United States there needs to be a more focused attempt at treating post-operative pain without use of opioids. Given the manipulation of soft tissue during a total knee arthroplasty there seems to be a high correlation with pain and myofascial pain syndrome. This study will include an experimental (trigger point injection) and control (sham injection) group who are all undergoing a total knee arthroplasty. This is a pilot study that will include a maximum of 100 total patients (although it is planned for the study to be much smaller with a planned 10-15 patients per group). The procedure that will be completed is a trigger point injection with use of 1% lidocaine without epinephrine along the distal aspect of the vastus medialis and lateralis, proximal aspect of the medial and lateral gastrocnemius muscle bellies. The sham injection will be completed by pressing the needle against the skin without injecting any fluid. There will be a "blind" between the patient and the needle with both arms of the study. These patients will be followed up on POD1, and during weeks 2 and 6 follow-up where they will be given questionnaires to assess pain (visual analogue scale) and opioid use, and asked to bring their opioid medications to the clinic to assess the morphine milligrams equivalent (MME).

ELIGIBILITY:
Inclusion Criteria:

* Aged 45 years or older
* Planned to undergo primary total knee arthroplasty
* Able to speak, read, and understand English
* Willing to complete a study questionnaires
* Willing to bring in their medications to be counted
* DoD beneficiaries
* No allergy to lidocaine
* Not fearful of needles.

Exclusion Criteria:

* Chronic opioid users (daily use of prescribed opioids for at least 90 days)
* Diagnosed with Fibromyalgia
* Non-English speaking
* Unable to read English
* Unable to understand English
* Pregnant
* Allergy to lidocaine
* Not willing to complete study questionnaires
* Not willing to bring in their medications to be counted
* Not a DoD beneficiary
* Fearful of needles

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2025-05-30 (Actual); Primary Completion 2025-08-25 (Actual); Study Completion 2025-08-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dustin L Bennett, Principal Investigator — David Grant
Locations (1):
- David Grant Medical Center, Fairfield, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental Group - Participants Receiving Trigger Point Injections | Sham Comparator - Participants Not Receiving Trigger Point Injections
Started | 6 | 5
Post Operative Day (POD) 1 | 6 | 5
Week 2 | 6 | 5
Week 6 | 3 | 3
Completed | 3 | 3
Not Completed | 3 | 2
Not completed — Limited timeline for follow-up restricted total number of participants for the last follow-up interv | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Group - Participants Receiving Trigger Point Injections | Sham Comparator - Participants Not Receiving Trigger Point Injections | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Categorical [Count of Participants; unit: Participants] — Population: Due to the total knee replacements not being conducted on 18 year olds or younger this demographic was not considered in our research
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 2 | 1 | 3
    >=65 years | 4 | 4 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 5 | 3 | 8
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.07 (2.15) | 33.84 (4.29) | 30.96 (3.22)
Number of Participants who are Military Retired or Military Dependents [Count of Participants; unit: Participants]
  Dependents | 1 | 2 | 3
  Retired | 5 | 3 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Pain Scores on the Visual Analog Scale
Description: 1. Change in Visual Analog Scale (VAS) pain scores
  The VAS is a numbered scale assessing pain severity using a number which describes the average level of pain since being discharged. Participants are to put a hash mark "/" on a numbered scale ranging from 0-100. Zero (0) is no pain and 100 is severe intolerable pain
Time Frame: From enrollment to the end of treatment at 6 weeks
Population: Limited timeline for follow-up restricted total number of participants for the last follow-up interval (6 week)
Measure: Mean (Standard Deviation); unit: Pain Scores on the Visual Analog Scale
Arm/Group | Experimental Group - Participants Receiving Trigger Point Injections | Sham Comparator - Participants Not Receiving Trigger Point Injections
Number analyzed (Participants) | 6 | 5
Pain Scores on the Visual Analog Scale
  Change from Baseline to Post Operative Day (POD) 1 | 51 (29.51) | 55 (22.64)
  Change from POD1 to week 2 follow-up | 40 (14.49) | 42 (24.9)
  Change from week 2 to week 6 follow-up: number analyzed (Participants) | 3 | 3
  Change from week 2 to week 6 follow-up | 30 (32.79) | 28.33 (18.93)

2. Secondary Outcome: Opioid Use
Description: 1. Compare the total opioid use between study groups (experimental, sham comparator).
  Opioid use will be measured during their inpatient stay using the Medication Administration Record (MAR) Summary in the electronic medical record; and completing an Opioid Use questionnaire and counting the number of pills remaining during post-operative/follow-up study visits. Inpatient opioid use will be calculated by using the morphine dosage and number of doses per day. Outpatient opioid use will be obtained by reviewing responses to the Opioid Use questionnaire and counting the number of pills remaining from the prescription given at the time of discharge. Participants will be asked to bring their medication (opioids) to their post-operative/follow-up study visits. This method will allow the investigator to measure total opioid use (injectable and pill) during their inpatient and outpatient course.
Time Frame: From enrollment to the end of treatment at 6 weeks
Population: Due to time constraints our study was only able to evaluate 3 participants in each arm of the study on the 6 week post-operative appointment.
Measure: Mean (Standard Deviation); unit: MME
Arm/Group | Experimental Group - Participants Receiving Trigger Point Injections | Sham Comparator - Participants Not Receiving Trigger Point Injections
Number analyzed (Participants) | 6 | 5
MME
  POD1 | 50.08 (36.89) | 68.60 (33.8)
  week 2 | 23.09 (12.21) | 19.09 (16.69)
  week 6: number analyzed (Participants) | 3 | 3
  week 6 | 1.33 (2.1) | 0 (0)

ADVERSE EVENTS:
Time Frame: from enrollment until the 6 week post-operative follow-up
Arm/Group | Experimental Group - Participants Receiving Trigger Point Injections | Sham Comparator - Participants Not Receiving Trigger Point Injections
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 0/6 | 0/5

LIMITATIONS AND CAVEATS:
Convenience sampling, Hawthorne effect, Sample Size, Peri-articular musculature targeted, Generalizability

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-04-23): https://cdn.clinicaltrials.gov/large-docs/23/NCT06955923/Prot_SAP_002.pdf
  • Informed Consent Form (2025-04-24): https://cdn.clinicaltrials.gov/large-docs/23/NCT06955923/ICF_001.pdf